CLINICAL TRIAL: NCT05985941
Title: Prospective Multi-omics Observational Study of Gynecological Rare Pathological Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-110-A
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Rare Gynecological Tumors; Multi-omics Analysis
Keywords: Genomics; Transcriptome; proteomics; metabonomics; Pathological omics; Imaging omics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to draw the characteristic maps of genomics, transcriptome, proteomics, metabolomics, etc. in 600 patients with gynecological rare pathological types of malignant tumors. Then it is planned to explore the molecular mechanism and find some new targets for diagnosis and treatment, and design and establish the database system of the above rare tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1)Pathological diagnosis: clear cell carcinoma (ovary, uterus), nerve small-cell carcinoma (ovary, uterus), carcinosarcoma or sarcoma (ovary, uterus), cervical gastric adenocarcinoma, ovarian germ cell tumor, ovarian sex cord stromal tumor, trophoblastic tumor, perivascular epithelioid cell tumor (PECOMA) and other rare gynecological tumors; 2)Received pathological results from tumor surgery; 3)The patient voluntarily participated in this research project with good compliance and was able to complete the enrollment according to the experimental requirements; 4)Sign the informed consent form and consent to the collection and use of their data, and consent to genomics, transcriptome and other tests.

Exclusion Criteria:

* 1)Patients with malignant tumors in other parts of the body; 2)Suffering from uncontrollable neurological diseases, psychiatric diseases, or psychiatric disorders; 3)Poor compliance and inability to cooperate and describe treatment responders.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rare gynecological tumors who underwent surgery in three hospitals, including Renji Hospital affiliated to Shanghai Jiaotong University School of Medicine, Sun Yat-sen Memorial Hospital affiliated to Sun Yat-sen University and the First Affiliated Hospital of University of Science and Technology of China, were diagnosed as clear cell carcinoma (ovary, uterus), neural small-cell carcinoma (ovary, uterus), carcinosarcoma or sarcoma (ovary, uterus), cervical gastric adenocarcinoma, ovarian germ cell tumor, ovarian sex cord stromal tumors, trophoblastic tumors, or perivascular epithelioid cell tumors (PECOMA), among others.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Multi-omics feature map | August 2023 to May 2028
  Draw the characteristic maps of imaging omics, genomics, transcriptome, proteomics, pathological omics, metabolomics, etc. of patients with gynecological rare pathological types of malignant tumors, and explore the molecular mechanism thus finding some new targets for diagnosis and treatment.
Database system | August 2023 to May 2028
  Design and establish the database system of the above gynecological rare pathological types of tumors.

SECONDARY OUTCOMES:
Correlation analysis | August 2023 to May 2028
  Integrate the characteristic maps of imaging omics, genomics, transcriptome, proteomics, pathological omics, metabonomics, etc. to study their possible relevance.